CLINICAL TRIAL: NCT02372539
Title: Pilot Project to Evaluate Hyperglycemia and Glucose Variability in Cancer Patients Receiving Dexamethasone
Brief Title: Glucose Variability in Cancer Patients Receiving Dexamethasone
Status: Withdrawn | Type: Observational
Why Stopped: COVID prevented accruals
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Society of Health-System Pharmacists (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1764.cc
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Hyperglycemia; Cancer
Keywords: dexamethasone
MeSH Terms: conditions — Hyperglycemia; Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-diabetes: Patients without diabetes will serve as the control group
  Interventions: Other: Control Group
- Diabetes: Patients with diabetes will be further stratified based upon antihyperglycemic medications (insulin versus oral medications)
  Interventions: Other: Diabetes

INTERVENTIONS:
Other: Diabetes — All patients enrolled in study will be given dexamethasone for prophylaxis of chemotherapy-induced nausea and vomiting. This will already be a part of their chemotherapy regimen and will not be prescribed by study investigators
  Groups: Diabetes
Other: Control Group — All patients enrolled in study will be given dexamethasone for prophylaxis of chemotherapy-induced nausea and vomiting. This will already be a part of their chemotherapy regimen and will not be prescribed by study investigators
  Groups: Non-diabetes

SUMMARY:
Dexamethasone is a steroid commonly used for the prevention of chemotherapy-induced nausea and vomiting (CINV). While effective, high dose dexamethasone is associated with numerous side effects, even when used for a short duration. One such effect is elevated blood glucose, or hyperglycemia. Current literature suggests increased risk of infection, poor wound healing, and increased mortality in non-cancer surgical patients with steroid-induced hyperglycemia. There is also evidence to support that elevations in blood glucose are associated with worsened outcomes in cancer patients. Much of this data comes from cancer patients that are treated in an inpatient setting where blood glucose is routinely checked. Limited data is available describing the fluctuations in blood glucose following dexamethasone administration in cancer patients being managed in an outpatient setting, such as the Anschutz Cancer Pavilion (ACP) Infusion Clinic. This study aims to characterize the effects dexamethasone has on blood glucose in cancer patients by utilizing Continuous Glucose Monitoring (CGM) devices. These devices are minimally invasive, are FDA approved, and can produce real-time data of blood glucose fluctuations over a course of 3-7 days. By inserting the devices under the skin of the abdomen, the investigators can evaluate the temporal relationship between glucose abnormalities and dexamethasone administration. Results from this study will not only increase the knowledge base of dexamethasone-induced hyperglycemia and identify patients at increased risk, but also allow future research to be conducted in order to determine if standard protocols can proactively minimize steroid-induced glucose fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant adult patients
* between 18-75 years of age
* are seen in the UCH outpatient cancer clinics for management of solid tumor and/or non-leukemia malignancies
* are prescribed high dose dexamethasone for CINV for no longer than 5 days, and
* have an absolute neutrophil count (ANC) > 1,500/mm3 and platelet count > 100,000/mm3 at time of glucose sensor placement.
* ANC of 1,500/mm3 is standard criteria for receiving outpatient chemotherapy.

Exclusion Criteria:

* leukemia-type malignancy
* require inpatient administration of chemotherapy
* are receiving chronic steroids
* have an ECOG/WHO/Zubrod score of 3 or 4
* have an ANC < 1,500 cells/mm3 at time of CGM device placement or are anticipated to have a decrease in ANC < 1,500 cells/mm3 during 5 days after sensor placement,
* have an active infection, or have significant cognitive impairment limiting their ability to use the CGM or complete a take-home diary.
* to further minimize the potential for infection, patients receiving chemotherapy regimens associated with a high (>20%) risk of febrile neutropenia, according to the 2014 NCCN guidelines, will also be excluded from study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with and without diabetes who are receiving intermittent high dose dexamethasone for prevention of chemotherapy-induced nausea and vomiting
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Hyperglycemic potential of dexamethasone | 7 days
  Determine the hyperglycemic potential associated with dexamethasone in cancer patients with and without diabetes.

SECONDARY OUTCOMES:
Measures of glucose variability | 7 days
  Evaluate measures of glucose variability including SD, percent coefficient of variance (%CV), high blood glucose index, and mean amplitude of glucose excursions (MAGE) in cancer patients receiving high dose dexamethasone for CINV prophylaxis
Time in hyperglycemia | 7 days
  Evaluate the time spent in hyperglycemic ranges (>180mg/dl) related to the time of dexamethasone administration
Hyperglycemia impact | 7 days
  Evaluate the impact of hyperglycemia on differences in clinical outcomes including patient reported adverse events and the incidence of those requiring medical intervention
Risk factors for hyperglycemia | 7 days
  Evaluate participant baseline characteristics to determine if risk factors for blood glucose elevations can be identified
Comparison of insulin versus oral antihyperglycemic medications | 7 days
  Evaluate if diabetes patients on oral medications versus insulin therapy demonstrate differences in blood glucose variability

CONTACTS AND LOCATIONS:
Overall Officials: Cindy O'Bryant, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States